CLINICAL TRIAL: NCT01200225
Title: Prospective Observational Study to Asses the Insulin Resistance (IR) and Its Impact on Sustained Virological Response in a Cohort of HCV-infected Patients Treated With Pegasys and Copegus
Brief Title: An Observational Study on The Impact of Insulin Resistance on Sustained Virological Response in Patients With Hepatitis C Treated With Pegasys (Peginterferon Alfa-2a) and Copegus (Ribavirin)
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML22790
Record Dates: First submitted 2010-09-10; First posted 2010-09-13 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Hepatitis C, Chronic
MeSH Terms: conditions — Hepatitis C, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Cohort

SUMMARY:
This prospective observational study will assess the insulin resistance and its impact on sustained virological response in patients with hepatitis C treated with Pegasys and Copegus. Data will be collected from each patient during the up to 72 weeks of treatment and for 24 weeks of treatment-free follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >/= 18 years of age
* Chronic hepatitis C (detectable HCV RNA)
* Initiation of treatment with Pegasys and Copegus

Exclusion Criteria:

* Participation in a clinical trial during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with inadequate response or intolerant to DMARDs and anti-TNF
Sampling Method: Probability Sample
Enrollment: 1155 (Actual)
Dates: Start 2010-02; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Effect of insulin resistance, defined as HOMA index > 2, on sustained virological response (HCV RNA assessed by Polymerase Chain Reaction assay) | 42 months

SECONDARY OUTCOMES:
Host-, virus- and treatment-related factors influencing virological response and sustained virological response | 42 months
Parameters of metabolic syndrome | 42 months
Management of insulin resistance | 42 months
Quality of life: Hepatitis Quality of Life Questionnaire (HQLQ) | 42 months
Safety: Incidence of adverse events | 42 months
Patient characteristics | 42 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Neuilly-sur-Seine, France